CLINICAL TRIAL: NCT01182922
Title: Is the Information About a Doctor or Possibility of Choosing Doctor's Gender Associated With Attendance to Screening Colonoscopy: Randomized Study With Three Types of Invitations.
Brief Title: Information About a Doctor or a Possibility of Choosing Doctor's Gender and Attendance to Screening Colonoscopy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CO-I
Record Dates: First submitted 2010-08-15; First posted 2010-08-17 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Colorectal Cancer; Screening
Keywords: Attendance; Colorectal cancer; Screening; Invitation letter
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Doctor's Information Invitation (Active Comparator): Standard invitation with additional leaflet containing information concerning particular doctor performing the examination, that is: his personal data (name, surname, academic title, workplace, picture) and data concerning experience and achievements of the center where he is employed.
  Interventions: Behavioral: Invitation letter
- Gender Preference Invitation (Active Comparator): Standard invitation with additional information about possibility of choosing doctor's gender, mentioned below proposed date of examination
  Interventions: Behavioral: Invitation letter
- Standard Invitation (Active Comparator): Standard invitation without additional information about a doctor or possibility of choosing doctor's gender.
  Interventions: Behavioral: Invitation letter

INTERVENTIONS:
Behavioral: Invitation letter — Invitation letter sent 6 weeks prior to prespecified screening colonoscopy appointment date and followed by reminder letter within 3 weeks if no response is received.

SUMMARY:
The purpose of the study is to investigate whether the information about a doctor or possibility to choose doctor's gender included in invitation letter is associated with attendance rate to screening colonoscopy.

DETAILED DESCRIPTION:
Study is performed as a part of NordICC (Clinical trials NCT 00883792) trial, which is intended to investigate the effect of screening colonoscopy on colorectal cancer incidence and mortality. NordICC trial is a multicenter, randomized study conducted in Norway, Sweden, Netherlands and Poland.

This study is designed to assess two factors potentially influencing patients attendance. These two factors are: identification of particular doctor performing examination and the possibility of choosing doctor's gender.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 55-64 years of age randomized to the screening arm of the NordICC trial in Poland

Exclusion Criteria:

* previous open colorectal surgery
* need for long term attention and nursing services (somatic or psychosocial reasons, mental retardation)
* ongoing cytotoxic treatment or radiotherapy for malignant disease
* severe chronic cardiac or pulmonary disease (NYHA III and IV)
* lifelong anticoagulant treatment
* coronary or cerebrovascular incident requiring hospitalization during the last three months
* residence abroad
* return of unopened letter of invitation and/or reminder, or message of death of the subject (not updated in Population Registry)
* failure to provide written informed consent
* screening colonoscopy within 10 years

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5100 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Percentage of invitees attending screening colonoscopy in each invitation letter group | 3 months from the primary assigned screening appointment date

SECONDARY OUTCOMES:
Percentage of forms with consent for examination, sent back after invitation letter but before reminding letter. Differences in attendance between men and women depending on type of the invitation. | 3 weeks after the date of invitation letter

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Regula, MD, PhD, Study Director — Center of Oncology Institute; Krzysztof Skoczylas, MD, Principal Investigator — Center of Oncology Institute; Michal F Kaminski, MD, Study Chair — Center of Oncology Institute
Locations (1):
- The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology,, Warsaw, Poland